CLINICAL TRIAL: NCT00198562
Title: Hypertension Control Based on Home Systolic Pressure Study (HOSP Study)
Brief Title: Hypertension Control Based on Home Blood Pressure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Collaborators: Japan Cardiovascular Research Foundation (Other)
Responsible Party: Yuhei Kawano, M.D., Ph.D., Director of Division of Hypertension and Nephrology, National Cardiovascular Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H16-CV-001; 200400510B
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Hypertension
Keywords: Antihypertensive therapy; Home blood pressure; Systolic blood pressure; Morning blood pressure; Calcium antagonist; Angiotensin receptor antagonist
MeSH Terms: conditions — Hypertension | interventions — amlodipine-losartan drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): target morning home blood pressure (below 130 mmHg vs 130-139 mmHg)
  Interventions: Drug: Amlodipine, Losartan
- 2 (Active Comparator): antihypertensive drug (amlodipine vs losartan)
  Interventions: Drug: Amlodipine, Losartan

INTERVENTIONS:
Drug: Amlodipine, Losartan — amlodipine: 2.5-10 mg once daily for 5 years losartan: 25-100 mg once daily for 5 years
  Other Names: other antihypertensive drugs (if required)

SUMMARY:
The aim of this trial is to study the effects of antihypertensive therapy based on home systolic blood pressure (BP) with different target levels using two classes of drugs.

The HOSP study is a multicenter, prospective, randomized, open, blinded endpoint study. The study subjects are 40-79 years old hypertensive patients. After a 4 weeks of baseline period, subjects are randomly assigned to (1) modest control group (morning home BP <140 mmHg) or (2) strict control group (morning home BP <130 mmHg), and to (a) amlodipine group or (b) losartan group. Additional antihypertensive drugs can be used if home BP is not controlled. Home BP is measured in the early morning and late evening. The participants will be followed up for 5 years.

DETAILED DESCRIPTION:
The aim of this trial is to study the effects of antihypertensive therapy based on home systolic blood pressure (BP) with different target levels using two classes of drugs.

The HOSP study is a multicenter, prospective, randomized, open, blinded endpoint study. Inclusion criteria are 40-79 years old treated or untreated hypertensive patients without serious medical conditions. After a 4 weeks of baseline period, subjects are randomly assigned to (1) modest control group (target morning home BP <140 mmHg) or (2) strict control group (morning home BP <130 mmHg), and to (a) amlodipine group (2.5-5 mg od) or (b) losartan group (25-50 mg od). Additional antihypertensive drugs (diuretics, beta-blockers and alpha-blockers) can be used if home BP is not controlled. Home BP is measured in the early morning and late evening. Primary end point is combined cardiovascular events.The participants will be followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension

Exclusion Criteria:

* Severe hypertension (treated with 3 or more antihypertensive drugs)
* Unable to change antihypertensive drugs to a calcium antagonist or an angiotensin antagonist
* Serious medical conditions
* Women who may become to be pregnant

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2000-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Combined cardiovascular events | 5 years

SECONDARY OUTCOMES:
Total mortality | 5 years
Cardiovascular mortality | 5 years
Myocardial infarction and new-onset angina | 5 years
Stroke and transient ischemic attack | 5 years
Renal failure | 5 years
Aortic and peripheral artery diseases | 5 years
Left ventricular mass and function | 5 years
Urinary albumin and renal function | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuhei Kawano, M.D., Ph.D., Principal Investigator — Division of Hypertension and Nephrology, National Cardiovascular Center
Locations (1):
- National Cardiovascular Center, Suita, Osaka, Japan